CLINICAL TRIAL: NCT02984345
Title: Does the Ingestion of Mycoprotein Elicit an Optimal Anabolic Response in Resting and Exercised Skeletal Muscle?
Acronym: ARM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 660065600
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mycoprotein beverage (Active Comparator)
  Interventions: Other: Mycoprotein beverage
- Milk protein beverage (Placebo Comparator)
  Interventions: Other: Milk protein beverage

INTERVENTIONS:
Other: Mycoprotein beverage — Mycoprotein protein beverage
  Arms: Mycoprotein beverage
Other: Milk protein beverage — Milk protein beverage
  Arms: Milk protein beverage

SUMMARY:
The present study will seek to quantify the muscle protein synthetic response to mycoprotein feeding, comparing it to milk protein as a gold standard and heavily researched positive control

ELIGIBILITY:
Inclusion Criteria:

• BMI between 18 and 30 -

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes)
* Any diagnosed cardiovascular disease or hypertension.
* Elevated blood pressure at the time of screening (e.g. blood pressure of ≥140/90mmHg).
* Chronic use of any prescribed or over the counter pharmaceuticals.
* A personal or family history of epilepsy, seizures or schizophrenia.
* Anyone with previous motor disorders.
* An allergy to mycoprotein / Quorn, penicillin, or milk.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Muscle fractional synthetic rate (muscle protein synthesis) | 7.5 hours

SECONDARY OUTCOMES:
Plasma amino acid concentration | 7.5 hours
Serum insulin concentration | 7.5 hours
Molecular markers of muscle anabolism | 7.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Exeter, Sports & Health Sciences, College of Life & Environmental Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No